CLINICAL TRIAL: NCT05218512
Title: Acute Effects of Whole-body Electromyostimulation on Energy Expenditure at Resting and During Uphill Walking in Healthy Young Men
Brief Title: WB-EMS Increase Energy Expenditure at Rest and During Uphill Walking Exercise
Status: Completed | Type: Observational
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Proffesor, Universidad de Granada
Other Study IDs: Impulse frequencies at rest
Record Dates: First submitted 2021-12-14; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Sports Physical Therapy
Keywords: Electrical stimulation; Energy expenditure; Obesity; Impulse intensities; Impulse frequencies
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- WB-EMS: Young recreationally active males without any disease.
  Interventions: Other: WB-EMS

INTERVENTIONS:
Other: WB-EMS — The group has been submitted to 2 experimental conditions:
  1. At rest with superimposed WB-EMS.
  2. During uphill walking exercise with superimposed WB-EMS.

SUMMARY:
Whole-body electrical stimulation (WB-EMS) has become increasingly popular as a tool to provide additional benefits compared to conventional exercise. However, the effects of the different electrical parameters on energy expenditure (EE) and respiratory exchange ratio (RER) remain poorly understood. This study aims to determine and compare the effects of different electrical frequencies applied with WB-EMS in EE and RER at supine resting and during uphill walking exercise

DETAILED DESCRIPTION:
Obesity is a critical public health problem worldwide since it is a risk factor for cardiovascular diseases and mortality. Increased body weight and obesity are the results of an imbalance between energy intake and energy expenditure (EE). Body weight regulation and obesity are highly influenced by different factors such as genetic, physiology, and socioeconomics. It is well known that physical exercise is an effective strategy to increase EE, improve body composition, physical fitness, and cardiometabolic risk factors. Unfortunately, the principal barriers to abstaining from exercise are time constraints, the risk of injuries, and the lack of enthusiasm observed during the exercise sessions. In this context, whole-body electromyostimulation (WB-EMS) training is becoming increasingly popular worldwide as a potential and attractive alternative to traditional training methods to increase EE. The present study aimed to determine and compare the effects of different electrical frequencies applied with WB-EMS in EE and RER at supine resting and during uphill walking exercise.

ELIGIBILITY:
Inclusion Criteria:

* (i) no previous experience with WB-EMS training
* (ii) having a stable body weight (variation of <5 kg in body weight over the previous 3 months)
* (iii) normal weight (body mass index (BMI) between 18.5-25.0 kg/m2)

Exclusion Criteria:

* (i) Suffering from any health problem that might be aggravated by exercise or any contraindications for WB-EMS, such as total endoprosthesis, epilepsy and abdomen/groin hernia
* (ii) Taking medications
* (iii) Chronic metabolic disease or cancer

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only males are recruited because we do not know if the period could affect to our results.
Study Population: We chose recreationally active males without any disease.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | It will be continuously measured through the entire test (60 minutes) of electromyostimulation with different impulse frequencies and intensities.
  Change in energy expenditure (kcal/min) by indirect calorimetry (Vyntus CPX Metabolic Cart)
Resting exchange ratio | It will be continuously measured through the entire test (60 minutes) of electromyostimulation with different impulse frequencies and intensities.
  Change in resting exchange ratio (kcal/min) by indirect calorimetry (Vyntus CPX Metabolic Cart)

SECONDARY OUTCOMES:
Pain perception | It will be measured at timepoints after the administration of each impulse frequency and before and after the whole application of electromyostimulation.
  Change in pain perception in different body structures by Visual Analogue Scales.
Impulse intensities | It will be measured with at timepoints after the administration of each impulse frequency.
  Change in impulse intensities in different body structures by whole-body electromyostimulation device.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Results will be shared with the scientific community.